CLINICAL TRIAL: NCT04851977
Title: A Phase I, First in Human (FIH), Randomised, Double-blind, Placebo-controlled, Dose-escalation Study to Evaluate Safety, Reactogenicity and Immunogenicity of the Recombinant Respiratory Syncytial Virus Vaccines (BARS13) When Administered Intramuscularly (IM) to Healthy Adult Volunteers
Brief Title: A First in Human Study to Evaluate the Safety and Immune Response to a Vaccine for the Treatment of a Respiratory Virus, When Administered Into the Arm in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Advaccine (Suzhou) Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ADVA-BARS13-001
Record Dates: First submitted 2021-04-13; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus (RSV); BARS13; Vaccines; Virus Diseases
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Virus Diseases

STUDY DESIGN:
Intervention Model Description: A total of up to 60 eligible participants will be enrolled and randomised in a 4:1 ratio (investigational vaccine versus placebo) to receive one of the following treatments:
  * BARS13 low dose (one dose of 10 μg rRSV-G protein/10 μg CsA by IM injection to the deltoid region of one arm, and one dose of placebo [saline/mannitol] by IM injection to the deltoid region of the other arm, given sequentially).
  * BARS13 high dose (IM injection of 10 μg rRSV-G protein/10 μg CsA administered to the deltoid region of each arm [one injection of 10 μg rRSV-G protein/10 μg CsA per arm], given sequentially). The high dose is twice the strength of the low dose.
  * Placebo (IM injection of saline/mannitol administered to the deltoid region of each arm [one injection per arm], given sequentially).
Who Masked: Participant, Investigator
Masking Description: This study is double-blinded. Sealed participant-specific code break envelopes will be produced by the unblinded statistician so that the treatment assigned to each participant can be obtained if required, in an emergency only, where knowledge of the randomisation code is required to provide appropriate treatment. The code break envelopes will be retained at the clinical unit in a secure, accessible location. Those blinded to study drug assignment include the sponsor, the PI, clinical study personnel participating in participants' care or clinical evaluations, and the study participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: low dose (Experimental): IM injection on Day 0 (12 active, 3 placebo); with follow up at 7 days ± 1 day post vaccination and at Day 30 ± 5 days and a final follow up/end of study (EOS) teleconference assessment at Day 60 ± 5 days.
  Interventions: Biological: Respiratory Syncytial Vaccine
- Cohort 2: low dose (Placebo Comparator): IM injection on Day 0 and at Day 30 (12 active, 3 placebo) with follow up at 7 days post vaccination (Day 7 ± 1 day and Day 37 ± 1 day) and Day 60 ± 5 days and a final follow up/ EOS teleconference assessment at Day 90 ± 5 days.
  Interventions: Biological: Placebo
- Cohort 3: high dose (Experimental): IM injection on Day 0 (12 active, 3 placebo); with follow up at 7 days ± 1 day post vaccination and at Day 30 ± 5 days and a final follow up/end of study (EOS) teleconference assessment at Day 60 ± 5 days.
  Interventions: Biological: Respiratory Syncytial Vaccine
- Cohort 4: high dose (Placebo Comparator): IM injection on Day 0 (12 active, 3 placebo); with follow up at 7 days ± 1 day post vaccination and at Day 30 ± 5 days and a final follow up/end of study (EOS) teleconference assessment at Day 60 ± 5 days.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Respiratory Syncytial Vaccine — BARS13 low dose (one dose of 10 μg rRSV-G protein/10 μg CsA by IM injection to the deltoid region of one arm, and one dose of placebo [saline/mannitol] by IM injection to the deltoid region of the other arm, given sequentially).
  Other Names: BARS13
  Arms: Cohort 1: low dose
Biological: Respiratory Syncytial Vaccine — BARS13 high dose (IM injection of 10 μg rRSV-G protein/10 μg CsA administered to the deltoid region of each arm [one injection of 10 μg rRSV-G protein/10 μg CsA per arm], given sequentially). The high dose is twice the strength of the low dose.
  Other Names: BARS13
  Arms: Cohort 3: high dose
Biological: Placebo — Placebo (IM injection of saline/mannitol administered to the deltoid region of each arm [one injection per arm], given sequentially).
  Arms: Cohort 2: low dose; Cohort 4: high dose

SUMMARY:
Advanced Vaccine Laboratories Pty Ltd is developing a recombinant Respiratory Syncytial Virus (rRSV) vaccine for the protection of children (6 months to 5 years old) and the elderly from RSV infection. Human RSV infects nearly all children by the age of two years, and it is a leading cause of severe lower respiratory tract (LRT) disease in both paediatric and elderly populations as well as in individuals was immune system is profoundly compromised.

DETAILED DESCRIPTION:
Advanced Vaccine Laboratories Pty Ltd is developing a recombinant Respiratory Syncytial Virus (rRSV) vaccine for the protection of children (6 months to 5 years old) and the elderly from RSV infection. Human RSV infects nearly all children by the age of two years, and it is a leading cause of severe lower respiratory tract (LRT) disease in both paediatric and elderly populations as well as in individuals was immune system is profoundly compromised. The investigational product BARS13 has not previously been administered to human subjects. The purpose of this study is to evaluate the safety of, and how the body reacts to, BARS13 investigational vaccine when administered in the arm to healthy adult participants aged 18 to 45 years according to a single (at Day 0) or repeat (at Day 0 and Day 30) vaccination schedule, with follow-up occurring for 60 days after the last vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 1. A male or female aged 18-45 years (inclusive) at the time of the first vaccination.

  2. Able to communicate effectively with study personnel and is considered reliable, willing, and cooperative in terms of compliance with the protocol requirements.

  3. Written informed consent signed prior to undertaking any protocol related procedures.

  4. Haematology, clinical chemistry and urinalysis test results not deviating from the normal reference range by age and gender to a clinically relevant extent at screening.

  5. Males must be surgically sterile (>30 days since vasectomy with no viable sperm), abstinent or, if engaged in sexual relations with a person of child-bearing potential, the participant and his partner must use an acceptable, highly effective, contraceptive method from screening and for a period of at least 3 months after the last dose of study drug. Acceptable methods of contraception are the use of condoms and an effective contraceptive for the female partner that could include: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, or intrauterine contraception/device. The PI is to assess the adequacy of methods of contraception on a case-by-case basis.

  6. Women of child-bearing potential (WOCBP) must use highly effective contraceptive measures (failure rate of < 1% per year when used consistently and correctly) throughout the study and intend to continue use of contraception for at least 3 months following the last vaccination. Highly effective contraceptive measures could include: combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone releasing system, bilateral tubal occlusion, vasectomised partner, and sexual abstinence. The PI is to assess the adequacy of methods of contraception on a case-by-case basis.

  7. Participant in otherwise general good health based on medical history and physical examination, as determined by the PI.

Exclusion Criteria:

* 1. Presence of clinically significant medical history, unstable chronic or acute disease, or physical, or laboratory findings that, in the opinion of the PI may potentially increase the expected risk of exposure to the investigational vaccine, compromise the safety of the participant, or interfere with any aspect of study conduct or interpretation of results.

  2. Body Mass Index (BMI) great than or equal to 40 at screening. 3. Significant infection or other acute illness, including fever over 37.5°C/99.5°F on the day of randomisation.

  4. Birthmarks, tattoos, wound or other skin conditions over the deltoid region of both arms that, in the PI's opinion, could reasonably obscure and interfere with evaluation of local injection site reactions.

  5. Inadequate venous access to allow collection of blood samples. 6. Breastfeeding or pregnant as confirmed by a positive serum beta human chorionic gonadotropin (.-HCG) pregnancy test at screening or positive urine pregnancy test at subsequent clinic visits at time points as delineated in the study schedule.

  7. Received any prophylactic or therapeutic vaccine, or investigational drug, within 3 months of first vaccination, or anticipated in the follow up period defined for this study.

  8. History of severe allergy (requiring hospital care), severe reaction to any drug or prior vaccination, or any known or suspected allergies or sensitivities to any component of the investigational vaccine or placebo.

  9. Immunosuppression caused by disease (such as human immunodeficiency virus [HIV]) or medications, immunosuppressive therapy (such as long-term systemic corticosteroids therapy).

  10. History of hepatitis B or hepatitis C infection. 11. History of autoimmune disorder. 12. History of splenectomy or of condition affecting splenic function. 13. History of malignancy of any organ system (other than localised basal cell carcinoma of the skin), treated or untreated, within the past five years, regardless of whether there is evidence of local recurrence or metastases.

  14. History of any neurological disorders or seizures. 15. Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.

  16. Receipt of immunoglobulins or blood products within 3 months of first vaccination.

  17. Requirement for antipyretic or analgesic medication on a daily or every other day basis from randomisation through 72 hours after vaccination.

  18. History of alcohol or drug abuse or psychiatric disorder that in the opinion of the PI could affect the participants' safety or compliance with study.

  19. Positive urine drug screen at screening, or pre-vaccination for any drug of abuse unless there is an explanation acceptable to the PI (e.g. the participant stated in advance that they consumed a prescription or over the counter product which contained the detected drug) and/or the participant had a negative urine drug screen on retest by the pathology laboratory.

  20. A positive alcohol breathalyser test at screening or pre-vaccination. 21. Participant unwilling to abstain from blood donation during the course of the study, and/or participation in any research study involving blood sampling (more than 450 mL /unit of blood), or blood donation to the Australian Red Cross Blood Service (ARCBS) or other blood bank during the 2 months prior to the screening visit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-04-07 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Incidence of systemic reactions | 7 days post vaccination
  Incidence of the systemic reactions (fatigue, myalgia, malaise, fever, rigors, arthralgia, nausea, diarrhoea, light-headedness, dizziness, hypersensitivity and headache) assessed by patient reported AEs and diary card
Incidence of local reactions | 7 days post vaccination
  Incidence of the local reactions (pain, tenderness, erythema, swelling, other e.g. ulceration, scabs, redness, induration, ecchymosis, oedema, itching and paraesthesia) at the site of vaccination assessed by patient reported AEs and diary card
Occurrence of any AE during a 30-minute post-vaccination safety observation period | 30 minutes post vaccination on Day 0 and 30
  Occurrence of any AE during a 30-day follow-up period after each vaccination.
Occurrence of any AE during a 30-day follow-up period after each vaccination | 30 days post vaccination
  Occurrence of any AE during a 30-day follow-up period after each vaccination.
Occurrence of any Serious Adverse Event (SAE) form baseline (Day 0) to the last visit | 60 days post last vaccination
  Occurrence of any Serious Adverse Event (SAE) form baseline (Day 0) to the last visit
Occurrence of any clinical laboratory abnormalities (Toxicity grade > or = 1) form baseline (Day 0) to the last visit | 60 days post vaccination
  Occurrence of any clinical laboratory abnormalities (Toxicity grade > or = 1) form baseline (Day 0) to the last visit

SECONDARY OUTCOMES:
Humoral response to BARS13: IgG antibody titers (GMTs) measured by ELISA prior to vaccination (Day 0) and post vaccination at Day 30 (all cohorts) and at Day 60 (cohorts 2 and 4 only) | Pre-vaccination
  Corrected post-dose Geometric Mean Titers (GMTs) of IgG antibody against RSV-G
Humoral response to BARS13: IgG antibody titers (GMTs) measured by ELISA prior to vaccination (Day 0) and post vaccination at Day 30 (all cohorts) and at Day 60 (cohorts 2 and 4 only) | 30 day post each vaccination
  Corrected post-dose Geometric Mean Titers (GMTs) of IgG antibody against RSV-G
Humoral response to BARS13: IgG antibody titers (GMFRs) measured by ELISA prior to vaccination (Day 0) and post vaccination at Day 30 (all cohorts) and at Day 60 (cohorts 2 and 4 only) | Pre-vaccination
  Post-dose Geometric Mean Fold Rises (GMFRs) from baseline of IgG antibody against RSV-G.
Humoral response to BARS13: IgG antibody titers (GMFRs) measured by ELISA prior to vaccination (Day 0) and post vaccination at Day 30 (all cohorts) and at Day 60 (cohorts 2 and 4 only) | 30 day post each vaccination
  Post-dose Geometric Mean Fold Rises (GMFRs) from baseline of IgG antibody against RSV-G.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Snyder, MBBS, Principal Investigator — The Alfred
Locations (1):
- Advanced Vaccine Laboratories Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
The results of this clinical trial may be published or presented at scientific meetings. If this is foreseen, the Investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. The Sponsor will comply with the requirements for publication of clinical trial results.